CLINICAL TRIAL: NCT00714753
Title: Pilot Evaluation of High Dose-Rate Brachytherapy ± Image-Guided Intensity Modulated Hypofractionated External Radiotherapy for Localized Prostate Cancer
Brief Title: Internal Radiation Therapy With or Without External-Beam Radiation Therapy in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000600446; P30CA015083 (NIH); MC0652 (Other: Mayo Clinic Cancer Center); 08-001451 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-07-11; First posted 2008-07-14 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Group (Experimental): Protocol treatment consists of either two high dose-rate (HDR) brachytherapy implantation sessions or one HDR brachytherapy session followed by external beam radiotherapy (EBRT). Each HDR session consists of two 9.5Gy fractions. After the first HDR session of two fractions, patients express a preference for: (1) a second HDR brachytherapy implantation session, or (2) EBRT. The second HDR session or EBRT will begin 2-4 weeks after the first HDR brachytherapy session.
  Interventions: Radiation: brachytherapy; Radiation: hypofractionated radiation therapy; Radiation: image-guided radiation therapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Radiation: brachytherapy
Radiation: hypofractionated radiation therapy
Radiation: image-guided radiation therapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase II trial is studying the side effects of internal radiation therapy when given with or without external-beam radiation therapy and to see how well it works in treating patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the tolerability of 2 radiotherapeutic regimens (high dose-rate brachytherapy [HDR] with or without image-guided intensity-modulated hypofractionated external beam radiotherapy [EBRT]), as measured by the Common Terminology Criteria for Adverse Events (CTCAE v3.0), in patients with localized prostate cancer.

Secondary

* Identify any associations between dose-volume parameters for organs at risk and the rate and severity of genitourinary or gastrointestinal adverse events.
* Evaluate patient preference with regard to selection of a second treatment (a second HDR brachytherapy session or an EBRT session).
* Evaluate patient-reported health-related quality of life (HRQOL) as measured by validated HRQOL instruments for 5 years.
* Describe the probability of freedom from biochemical and clinical failure.
* Describe the probability of freedom from salvage androgen suppression.

OUTLINE: Patients undergo high dose-rate (HDR) brachytherapy (2 fractions ≥ 5 hours apart). Beginning 2-4 weeks after completion of the first HDR brachytherapy session, patients undergo either a second session of HDR brachytherapy (2 fractions ≥ 5 hours apart) OR image-guided intensity-modulated hypofractionated external beam radiotherapy once daily 5 days a week for 3 weeks.

Quality of life is assessed at baseline, prior to the second treatment session, at 1 and 6 months after completion of treatment, every 6 months for 3 years, and then annually for 2 years.

After completion of study treatment, patients are followed at 1 and 6 months, every 6 months for 3 years, and then annually for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate, meeting one of the following criteria:

  * Low-risk disease (T1-T2a, Gleason score ≤ 6, and PSA < 10 ng/mL)
  * Low intermediate-risk disease (T1-T2c, Gleason score ≤ 6, and PSA < 20 ng/mL OR T1-T2a, Gleason score 7, and PSA < 10 ng/mL)
* No known nodal (N0 or NX) or distant (M0 or MX) metastases
* No pubic arch interference, as defined by either of the following:

  * Maximum transrectal ultrasound-determined anterior-posterior (z-axis) dimension < 4.3 cm
  * No more than 25% prostate volume blocked (by pubic arch) on CT scan simulation at A10°I beam's eye view
* Prostate planimetry volume ≤ 60 cc as determined by step-section transrectal ultrasound
* American Urological Association voiding symptom index ≤ 12
* Peak uroflow rate (Q_max) ≥ 12 cc/second
* Post-void ultrasound bladder residual volume ≤ 100 cc

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Life expectancy ≥ 5 years
* WBC > 2,000/μL
* Platelet count > 100,000/μL
* PT < 1.5 times upper limit of normal
* No diabetes mellitus associated with vascular ulcers or wound-healing problems
* No blood dyscrasias
* No inflammatory bowel disease
* No connective tissue disorder
* No other prior or concurrent invasive malignancy (except nonmelanoma skin cancer) or lymphomatous or hematological malignancy (except chronic lymphocytic leukemia/lymphoma) unless patient has been continually disease-free for ≥ 5 years
* No medical or psychiatric condition that would preclude giving informed consent or complying with study treatment
* Able to undergo anesthesia

PRIOR CONCURRENT THERAPY:

* No prior transurethral resection of the prostate
* No prior prostatic cryoablation or high-intensity focused ultrasound
* No prior prostatectomy
* No prior prostatic enucleation
* No prior pelvic external beam radiotherapy
* No prior radionuclide prostate brachytherapy
* No prior hemi- or total hip arthroplasty
* Neoadjuvant androgen suppression therapy allowed provided it was initiated 2-6 months prior to study entry and its total duration is ≤ 6 months
* No concurrent anticoagulation therapy, including heparin or coumadin

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Pisansky, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (HDR ± EBRT): Protocol treatment consists of either two high dose-rate (HDR) brachytherapy implantation sessions or one HDR brachytherapy session followed by external beam radiotherapy (EBRT). Each HDR session consists of two 9.5Gy fractions. After the first HDR session of two fractions, patients express a preference for: (1) a second HDR brachytherapy implantation session, or (2) EBRT. The second HDR session or EBRT will begin 2-4 weeks after the first HDR brachytherapy session.
Period: Overall Study
Arm/Group | Arm 1 (HDR ± EBRT)
Started | 5
HDR Brachytherapy | 5
External Beam Radiotherapy (EBRT) | 1
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients who were eligible and began treatment. Only 1 patient was registered to the HDR+EBRT arm. Due to protected health information, listing only 1 patient's results is contraindicated.
Arm/Group | Arm 1 (HDR ± EBRT)
Number analyzed (Participants) | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.0 [65.0 to 72.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Treatment Tolerance (Genitourinary [GU] or Gastrointestinal [GI] Adverse Events)
Description: Separately evaluate the tolerance of 2 radiotherapeutic regimens (HDR alone and HDR followed by hypofractionated EBRT) using the Common Terminology Criteria for Adverse Events (CTCAE v3.0). The specific adverse events (AEs) are early (i.e., within 270 days of treatment completion) grade >3 genitourinary (GU) and/or gastrointestinal (GI) AEs, late grade 2 GU and GI AEs, and late grade ≥3 GU and GI AEs.
Time Frame: From baseline to 3 years after registration
Population: All patients registered to a dose escalation Phase I group were analyzed for this endpoint. Only 1 patient was registered to the HDR+EBRT arm. Due to protected health information, listing only 1 patient's results is contraindicated.
Measure: Number; unit: events
Arm/Group | Arm 1 (HDR ± EBRT)
Number analyzed (Participants) | 5
events | 3

2. Secondary Outcome: Association Between Dose-volume Limitations for Organs at Risk and Rate and Severity of GU or GI Adverse Events
Description: Dose-volume limitations for organs at risk will be analyzed byassociating GU or GI AEs (both rate and severity) with dosimetric parameters using simple correlational methods. These parameters will include (1) bladder V80, V60, V50, and Dmax; (2) penile bulb median dose; (3) rectum V80, V60, V50 and Dmax; and (4) urethra V120, V110, V100, and Dmax.
Time Frame: From baseline to 5 years after registration
Population: No patients registered to a dose escalation Phase I group were analyzed for this endpoint. With only 5 patients, the study team deemed that the information would be unsuitable.
Arm/Group | Arm 1 (HDR ± EBRT)
Number analyzed (Participants) | 0

3. Secondary Outcome: Patient Preference for a Second Treatment (a Second High Dose-rate Brachytherapy Session or an External Beam Radiotherapy Session)
Description: Patient preference for second treatment (group 1 or group 2) will be assessed using a Treatment Preference Questionnaire (Appendix IX) developed specifically for this study. Qualitative and quantitative analyses will be performed on patient responses to the questions posed after choosing their second treatment in an exploratory fashion.
Time Frame: From baseline until the end of the first treatment
Population: None of the enrolled patients were analyzed for this endpoint due to too few patients.
Arm/Group | Arm 1 (HDR ± EBRT)
Number analyzed (Participants) | 0

4. Secondary Outcome: Changes in Health-related Quality of Life Scores
Description: A pretest-posttest design will be employed to detect changes in HRQOL scores over time. The HRQOL scores will be calculated per assessment, as appropriate. Each construct will be standardized to a range of 0-100 so that comparison across constructs is facilitated. Sets of difference scores will be computed: 1) differences between baseline and treatment completion (at 1 month post treatment follow up), and 2) differences between treatment completion and all post-treatment follow-up examinations for up to five years after finishing the protocol treatment (see Section 4.1 for specific HRQOL instruments to be completed at follow-up visits). The first analysis will allow for determination of the short-term impact of treatment on HRQOL, while the second will investigate the long-term treatment effect. Student's t-test methodology will be applied to the differences at end of treatment (1 month post treatment follow up) and at each follow-up.
Time Frame: From baseline to 5 years after registration
Population: None of the enrolled patients were analyzed for this endpoint due to too few patients.
Arm/Group | Arm 1 (HDR ± EBRT)
Number analyzed (Participants) | 0

5. Secondary Outcome: Freedom From Biochemical and Clinical Failure
Description: Freedom from biochemical and clinical failure, will be analyzed using Kaplan-Meier procedures. Estimates will be drawn from the Kaplan-Meier curves for the probability of freedom from biochemical and clinical failure.
Time Frame: From baseline to 5 years after registration
Population: With only 5 patients, the study team deemed that the information would be unsuitable.
Arm/Group | Arm 1 (HDR ± EBRT)
Number analyzed (Participants) | 0

6. Secondary Outcome: Freedom From Salvage Androgen Suppression Treatment
Description: Estimates will be drawn from the Kaplan-Meier curves for the probability of freedom from salvage androgen suppression therapy.
Time Frame: From baseline to 5 years after registration
Population: With only 5 patients, the study team deemed that this information would be unsuitable.
Arm/Group | Arm 1 (HDR ± EBRT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed within 7 days of High Dose-Rate Radiation (HDR) and External beam radiation therapy (EBRT), and at one month after completion of therapy, 6 months after registration, then every 6 months x 5 (through year 3), then every 12 months for years 4-5, then off study. Up to 5 years.
Description: CTCAE term & grade: The descriptions & grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation & scientific analysis & is a single MedDRA Lowest Level Term (LLT). Only 1 patient was registered to the HDR+EBRT arm. Due to protected health information, listing only 1 patient's results is contraindicated.
Arm/Group | Arm 1 (HDR ± EBRT)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (HDR ± EBRT) (N=5)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (9)
Flatulence (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 2 (2)
Bladder pain (Renal and urinary disorders) | 1 (1)
Bladder stenosis (Renal and urinary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 3 (3)
Urethral hemorrhage (Renal and urinary disorders) | 2 (2)
Urethral pain (Renal and urinary disorders) | 4 (6)
Urinary frequency (Renal and urinary disorders) | 4 (12)
Urinary incontinence (Renal and urinary disorders) | 3 (5)
Urinary retention (Renal and urinary disorders) | 3 (5)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 4 (5)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Prostatic hemorrhage (Reproductive system and breast disorders) | 2 (2)
Prostatic pain (Reproductive system and breast disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes